CLINICAL TRIAL: NCT00527631
Title: Adjuvant Whole Abdominal Intensity Modulated Radiotherapy (IMRT) for High Risk Stage FIGO III Patients With Ovarian Cancer: Pilot Trial of a Phase I/II Study
Brief Title: Adjuvant Whole Abdominal Intensity Modulated Radiotherapy (IMRT) for High Risk Stage FIGO III Patients With Ovarian Cancer
Acronym: OVAR-IMRT-01
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 176/2005
Record Dates: First submitted 2007-09-07; First posted 2007-09-11 (Estimated); Last update posted 2007-09-11 (Estimated); Status verified 2007-08

CONDITIONS: Ovarian Cancer
Keywords: advanced ovarian cancer; whole abdominal irradiation; intensity modulated radiotherapy; ovarian cancer stage FIGO III
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: whole abdomen irradiation using IMRT — Whole abdomen irradiation as consolidation therapy using intensity modulated radiation therapy (IMRT) to a total dose of 30 Gy in 1.5 Gy fractions

SUMMARY:
The prognosis for patients with advanced epithelial ovarian cancer remains poor despite aggressive surgical resection and platinum-based chemotherapy. More than 60% of patients will develop recurrent disease, principally intraperitoneal, and die within 5 years. The use of whole abdominal irradiation (WAI) as consolidation therapy would appear to be a logical strategy, but despite whole abdominal irradiation has clinically proven efficacy the use of radiotherapy in ovarian cancer has profoundly decreased mainly due to high treatment-related toxicity. Modern intensity-modulated radiation therapy (IMRT) could allow to spare kidneys, liver, and bone marrow while still adequately covering the peritoneal cavity with a homogenous dose.

This study will evaluate feasibility and toxicity of adjuvant consolidation whole abdominal intensity modulated radiotherapy (IMRT) for high risk stage FIGO III patients with ovarian cancer.

DETAILED DESCRIPTION:
The prognosis for patients with advanced epithelial ovarian cancer remains poor despite aggressive surgical resection and platinum-based chemotherapy. More than 60% of patients will develop recurrent disease, principally intraperitoneal, and die within 5 years. The use of whole abdominal irradiation (WAI) as consolidation therapy would appear to be a logical strategy, but despite whole abdominal irradiation has clinically proven efficacy the use of radiotherapy in ovarian cancer has profoundly decreased mainly due to high treatment-related toxicity. Modern intensity-modulated radiation therapy (IMRT) could allow to spare kidneys, liver, and bone marrow while still adequately covering the peritoneal cavity with a homogenous dose.

The OVAR-IMRT-01 study is a single center pilot trial of a phase I/II study. Patients with advanced ovarian cancer stage FIGO III (R1 or R2< 1cm) after surgical resection and platinum-based chemotherapy will be treated with whole abdomen irradiation as consolidation therapy using intensity modulated radiation therapy (IMRT) to a total dose of 30 Gy in 1.5 Gy fractions. A total of 8 patients will be included in this trial. For treatment planning bone marrow, kidneys, liver, spinal cord, vertebral bodies and pelvic bones are defined as organs at risk. The planning target volume includes the entire peritoneal cavity plus pelvic and para-aortic node regions.

The primary endpoint of the study is the evaluation of the feasibility of intensity-modulated WAI, the secondary endpoint is evaluation of the toxicity of intensity modulated WAI before continuing with the phase I/II study. The aim is to explore the potential of IMRT as a new method for WAI to decrease the dose to kidneys, liver, bone marrow while covering the peritoneal cavity with a homogenous dose, and to implement whole abdominal intensity-modulated radiotherapy into the adjuvant multimodal treatment concept of advanced ovarian cancer FIGO stage III.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed ovarian cancer stage FIGO III
* grade 2 or 3
* maximal typical surgical resection (including at least total abdominal hysterectomy, bilateral adnexectomy, omentectomy, debulking of tumour masses)
* postoperative residual tumour of less than 1 cm (maximal diameter of largest tumour residual is 1 cm)
* adjuvant chemotherapy consisting of six courses of carboplatin/paclitaxel or carboplatin/docetaxel
* complete remission after chemotherapy
* Karnofsky performance Score >60
* patients > 18 and < 75 years of age
* written informed consent

Exclusion Criteria:

* stage FIGO I or II
* stage IV (distal metastasis)
* stage III R2 > 1 cm
* delayed wound healing post laparotomy
* neutrophil count (ANC) < 2000/ml before radiotherapy
* platelets < 100000/ml
* connective tissue disease, sclerodermia
* clinically active renal, hepatic, cardiac, metabolic, respiratory, coagulation or haematopoietic disease
* participation in another clinical trial
* patient refusal

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2006-07; Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
feasibility | 8 weeks

SECONDARY OUTCOMES:
toxicity | baseline, weekly during the 4 weeks of radiation. Follow up 6 weeks, 3 months, 6 months, 9 months, 12 months post treatment, and then every 6 months for 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Harms, MD, Principal Investigator — Heidelberg University
Locations (1):
- Department of Radiation Oncology, University of Heidelberg, Im Neuenheimer Feld 400, Heidelberg, Germany